CLINICAL TRIAL: NCT06891209
Title: Exploration of HRQOL and Urinary Outcomes Following Partial Cystectomy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vidit Sharma, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 23-007176; NCI-2025-00372 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-007176 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observational - Radical Cystectomy: Patients complete questionnaires and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Observational - Partial Cystectomy: Patients complete questionnaires and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study explores and compares health-related quality of life and urinary outcomes in postoperative partial cystectomy and matched radical cystectomy patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Explore and compare urinary outcomes in postoperative partial cystectomy patients and matched radical cystectomy patients through patient-filled questionnaires.

II. Explore and compare health related quality of life in postoperative partial cystectomy and matched radical cystectomy patients using patient-filled questionnaires.

III. Explore the relationship of patient-specific characteristics, ranging from demographic characteristics and clinicopathologic characteristics, on variation in HRQOL and urinary outcomes among the partial cystectomy and radical cystectomy cohorts.

OUTLINE: This is an observational study.

Patients complete questionnaires and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Currently living partial cystectomy patients in Mayo Urology's cystectomy registry and patients undergoing radical or partial cystectomy
* Matched 2:1 living radical cystectomy to partial cystectomy patients
* Either urothelial or non-urothelial histology

Exclusion Criteria:

* Partial cystectomy patients that underwent subsequent radical cystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Currently living partial cystectomy patients in Mayo Urology's cystectomy registry and patients undergoing radical or partial cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life - EORTC QLQ-C30 | Up to 1 year
  Assessed using the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30), which is designed to measure cancer patients' physical, psychological and social functions. It is a 30-item questionnaire related to symptoms and activities during the past week. Responses are recorded on a scale of 1-4 where 1=not at all, 2=a little, 3=quite a bit, and 4=very much. Scores among partial cystectomy patients will be compared to radical cystectomy patients.
Self-reported urinary outcomes | Up to 1 year
  Assessed using the EORTC Quality of Life Questionnaire - Muscle Invasive Bladder Cancer (EORTC QLQ-BLM30), a 30-item questionnaire related to general symptoms experienced during the past week or during the past 4 weeks. Responses are recorded on a scale of 1-4 where 1=not at all, 2=a little, 3=quite a bit, and 4=very much. Scores among partial cystectomy patients will be compared to radical cystectomy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vidit Sharma, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials